CLINICAL TRIAL: NCT03810976
Title: Open-label, Phase II Trial of Eribulin in Combination With Gemcitabine in Previously Treated Patients With Advanced Liposarcoma or Leiomyosarcoma
Brief Title: A Study of Eribulin With Gemcitabine in Patients With Advanced Liposarcoma or Leiomyosarcoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Principal Investigator, Hyo Song Kim, professor, Yonsei University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4-2017-0933
Record Dates: First submitted 2019-01-16; First posted 2019-01-22 (Actual); Last update posted 2022-06-16 (Actual); Status verified 2022-06

CONDITIONS: Sarcoma
MeSH Terms: conditions — Sarcoma | interventions — eribulin; Gemcitabine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- eribulin+gemcitabine (Experimental): The dose is 1.4 mg/m2 for 5 minutes intravenously. If necessary, the dose may be diluted in up to 100 mL of saline solution prior to intravenous administration. Gemcitabine doses 1000 mg/m2 intravenously for 30 minutes. After completion of the eribulin injection, intravenously inject gemcitabine. One cycle is 3 weeks, and the treatment is carried out on the 1st day and the 8th day for each cycle.
  Interventions: Drug: Eribulin, gemcitabine

INTERVENTIONS:
Drug: Eribulin, gemcitabine — Elibulin 1.4mg/m2 Intravenous for 5minutes. Day 1& Day 8 every 3 weeks Gemcitabine 1000mg/m2 intraveoust for 30 minutes, Day 1& Day 8 every 3 weeks

SUMMARY:
The eribulin, a microtubule-dynamics inhibitor was approved for specific subtypes of STS. Eribulin demonstrated significantly better OS compared to dacarbazine in previously treated patients with liposarcoma and leiomyosarcoma and approved as standard treatment. However, the median progression free survival (PFS) and response rate (RR) was similar for both groups which remains modest outcome of 2.6 months of PFS and 4% of RR. Therefore, to improve antitumor activity, further combination strategy is strongly warranted. Based on the previous studies, investigators suggest phase II trial of eribulin and gemcitabine combination in previously treated patients with unresectable, advanced, or metastatic leiomyosarcoma or liposarcoma.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed advanced liposarcoma or leiomyosarcoma with 1-2 prior chemotherapy including anthracycline (unless contraindicated)
2. ECOG performance status of 0-2
3. Measurable or evaluable disease (RECIST 1.1.)
4. Adequate laboratory findings

   * Hb ≥ 9.0 g/dL
   * Absolute neutrophil count ≥ 1000 /µL
   * Platelet ≥ 75,000/ µL
   * Total Bilirubin: ≤ 1.5 × UNL (upper normal limit) (≤ 2 × UNL in patients with liver metastasis)
   * Serum Creatinine: ≤1.5 X upper limit of normal (ULN) OR ≥ Creatinine Clearance 60 mL/min (Cockcroft-Gault) for patients with creatinine levels > 1.5 X institutional ULN
   * AST(SGOT)/ALT(SGPT): ≤ 3.0 × UNL or ≤ 5.0 × UNL (in patients with liver metastasis)
   * Alkaline Phosphatase : ≤ 3.0 × UNL or ≤ 5.0 × UNL (in patients with liver or bone metastasis)
   * Prothrombin time and partial thromboplastin time : ≤1.5 X ULN
5. Female patient of childbearing potential has a negative serum or urine pregnancy test within 72 hours prior

Exclusion Criteria:

1. More than 3 prior cytotoxic agents
2. Patient who has had chemotherapy, radiotherapy, or biological therapy within 2 weeks prior to entering the study
3. Uncontrolled or active CNS metastasis and/or carcinomatous meningitis
4. Patient has known hypersensitivity to the components of study drugs or its analogs.
5. Patient is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the study.
6. Long QT Syndrome ≥480 ms
7. peripheral neuropathy ≥2 with previous treatment
8. unstable cardiovascular disease
9. Symptomatic interstitial lung disease (ILD) or presence of ILD on chest X-ray

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2018-03-27 (Actual); Primary Completion 2022-05-30 (Actual); Study Completion 2022-05-30 (Actual)

PRIMARY OUTCOMES:
progression free survival | 12 weeks
  To evaluate antitumor efficacy of eribulin and gemcitabine combination

SECONDARY OUTCOMES:
adverse event | through study completion, an average of 6 months
  to evaluate safety

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Yonsei University Health System, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No